CLINICAL TRIAL: NCT02627209
Title: Non-infectious and Infectious Uveitis Diagnosis
Brief Title: The Serum Angiotensin Converting Enzyme and Lysozyme Levels in Patients Non-infectious and Infectious Uveitis
Acronym: uveitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ozlem Sahin (Other)
Responsible Party: Sponsor-Investigator, Ozlem Sahin, Medical Doctor, Specialist in Ophthalmology, Uveitis and Ocular Immunology, Dünyagöz Hospital
Organization: Dünyagöz Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DGH-070
Record Dates: First submitted 2015-11-26; First posted 2015-12-10 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Sarcoidosis; Tuberculosis
Keywords: Angiotensin converting enzyme; Lysozyme; Ankylosing spondylitis; Behcet's disease; Sarcoidosis; Syphilis; Tuberculosis; Ocular inflammation
MeSH Terms: conditions — Sarcoidosis; Tuberculosis; Spondylitis, Ankylosing; Behcet Syndrome; Syphilis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- serum angiotensin converting enzyme (Active Comparator): spectrophotometric assay
  Interventions: Other: spectrophotometric assay; Other: radial immunodiffusion
- serum lysozyme (Active Comparator): radial immunodiffusion
  Interventions: Other: spectrophotometric assay; Other: radial immunodiffusion

INTERVENTIONS:
Other: spectrophotometric assay — measurement of enzyme activity in the serum
Other: radial immunodiffusion — measurement of the precipitated ring diameters showing enzyme activity in the serum

SUMMARY:
This study evaluates the significance of differences in serum angiotensin converting enzyme and lysozyme levels of patients with ocular involvement of other autoimmune inflammatory and infectious diseases.

DETAILED DESCRIPTION:
Increased serum levels of angiotensin converting enzyme and lysozyme are considered as inflammatory markers for diagnosis of sarcoidosis which is an autoimmune inflammatory disease. Sarcoidosis, ankylosing spondylitis and Behcet's disease are the most common autoimmune inflammatory diseases involving the eye.

Elevated serum angiotensin converting enzyme levels have also been reported in tuberculosis. Syphilis and tuberculosis are the most common infectious diseases involving the eye.

ELIGIBILITY:
Inclusion Criteria:

* Subjects have ocular inflammation diagnosed as sarcoidosis, ankylosing spondylitis, behcet's disease
* Subjects have ocular infection diagnosed as tuberculosis and syphilis
* Subjects have refractive errors only

Exclusion Criteria:

* Subjects using ACE inhibitors, systemic steroids, immunosuppressive or immunomodulatory therapies

Ages: 9 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-02 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Analysis of serum angiotensin converting enzyme level | 1 day

SECONDARY OUTCOMES:
Analysis of serum lysozyme level | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Pallikaris, MD, Study Chair — DunyaGoz Hospital, Etiler, yanarsu sokak no.1 besiktaş Istanbul Turkey
Locations (1):
- DunyaGoz hospital Tunus caddesi no.28 kavaklidere, Çankaya, Ankara, Turkey (Türkiye)

REFERENCES:
- [Result] Birnbaum AD, Oh FS, Chakrabarti A, Tessler HH, Goldstein DA. Clinical features and diagnostic evaluation of biopsy-proven ocular sarcoidosis. Arch Ophthalmol. 2011 Apr;129(4):409-13. doi: 10.1001/archophthalmol.2011.52. PMID 21482866
- [Result] Sen DK, Sarin GS. Immunoassay of serum muramidase (lysozyme) in ocular diseases. Indian J Ophthalmol. 1987;35(5-6):103-7. PMID 3508756
- [Derived] Sahin O, Ziaei A, Karaismailoglu E, Taheri N. The serum angiotensin converting enzyme and lysozyme levels in patients with ocular involvement of autoimmune and infectious diseases. BMC Ophthalmol. 2016 Feb 16;16:19. doi: 10.1186/s12886-016-0194-4. PMID 26879979